CLINICAL TRIAL: NCT05726916
Title: Eculizumab in Hypertensive Emergency-associated Hemolytic Uremic Syndrome: a Randomized Multicenter Controlled Trial
Brief Title: Eculizumab in Hypertensive Emergency-associated Hemolytic Uremic Syndrome
Acronym: HYPERSHU
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP211039
Record Dates: First submitted 2022-12-16; First posted 2023-02-14 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-09

CONDITIONS: Hypertensive Emergency-associated Hemolytic Uremic Syndrome
Keywords: Eculizumab; Hypertensive emergency; atypical hemolytic uremic syndrome; complement; acute kidney injury; end stage renal disease
MeSH Terms: conditions — Hypertensive Crisis; Atypical Hemolytic Uremic Syndrome; Acute Kidney Injury; Kidney Failure, Chronic | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: The present proposal is a randomized, controlled, multicenter, open-labelled study.
  In the experimental group, Ecu will be administered at randomization according to usual recommendations in aHUS (4 intravenous administrations, 900mg/w until W4 then 1200mg/2w starting at W5, until W13).
  In both experimental and control group, BP control with systematic maximum tolerated dose of RAS blockers will be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Eculizumab IV administration (900mg/w during 4w then 1200 mg at w5 and 1200mg/2w for 8w) + Blood pressure control with renin angiotensin system blockers
  Interventions: Drug: Soliris®
- Control group (Active Comparator): Blood pressure control with renin angiotensin system blockers
  Interventions: Drug: Renin angiotensin system blockers

INTERVENTIONS:
Drug: Soliris® — Eculizumab IV administration (900mg/w during 4w then 1200 mg at w5 and 1200mg/2w for 8w) + Blood pressure control with renin angiotensin system blockers
  Other Names: Eculizumab
  Arms: Experimental group
Drug: Renin angiotensin system blockers — Blood pressure control with renin angiotensin system blockers
  Arms: Control group

SUMMARY:
Hemolytic and uremic syndrome (HUS) is a clinic-biological syndrome related to thrombotic microangiopathy affecting predominantly the kidney. Atypical HUS (aHUS) has been historically defined as HUS occurring in the absence of infectious event. The role of complement dysregulation in aHUS pathophysiology has been largely demonstrated, since C genetic rare variants are present in 60-70% aHUS patients. In line with the frequency of C dysregulation in aHUS, Eculizumab, an anti-C5 monoclonal antibody, has dramatically improved aHUS patients prognosis.

Numerous conditions have been associated with aHUS, including hypertensive emergency (HE), a syndrome of acute blood pressure flare associated with end-organ damage. In cases of HE-aHUS, whether primary aHUS is complicated by secondary HE, or primary HE leads to secondary aHUS is still debated.

The investigators recently demonstrated that C genetic variants frequency was similar in patients with HE-aHUS and patients with aHUS without HE, suggesting a major role for C dysregulation in HE-aHUS. Consequently, the investigators propose to evaluate, in HE-aHUS patients, the benefit of a strategy with early Eculizumab therapy (used within its marketing authorization and its conditions of refunding by the health insurance in usual care), compared to standard of care including tight blood pressure control.

The hypothesis suggests that C dysregulation may impact renal prognosis of HE-aHUS patients. The investigator's aim to demonstrate that early Eculizumab therapy improves prognosis of HE-aHUS patients.

Method

The HYPERSHU study is a randomized, controlled, open-labelled study including HE-aHUS patients with severe AKI and no evidence of other conditions associated with HUS (infections, autoimmunity, drugs, pregnancy). The investigators plan to include 62 patients. Patients will be randomized in 2 arms:

* Early Eculizumab therapy (for 3 months) added to standard of care (tight blood pressure control).
* Standard of care alone with tight blood pressure control. Renal function after 6 months is the primary evaluation criterium.

HE is a frequently associated with aHUS, and strongly impacts patient renal prognosis. Efficient therapeutic strategies are still lacking for this condition. The HYPERSHU study will allow to evaluate the benefit of early Eculizumab therapy in patients with HE-aHUS and severe renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18years
* Hospitalization for HE-aHUS within prior 10 days:

  * Presume acute renal failure (renal replacement therapy or serum creatinine ≥ 354µM)
  * Mechanical hemolysis including: anemia, thrombopenia, and: low haptoglobin (<LNL), or elevated LDH (>1,5UNL), or presence of schistocytes
  * Severe hypertension with systolic blood pressure >180mmHg or diastolic blood pressure>110mmHg
  * Target organ damage, including neurological involvement (notably hypertensive encephalopathy, headache, confusion, nausea, posterior reversible encephalopathy syndrome), or cardiovascular involvement (notably acute left ventricular failure, acute pulmonary edema, acute cardiac ischemia, chest pain, dyspnea, palpitations), or ophtalmological involvement (notably ischemic retinopathy or blurred vision)
* Effective contraception during the study and for at least 5 months after the last dose of treatment with eculizumab
* Subject affiliated to a social security regimen
* Subject having signed written informed consent.

Exclusion Criteria:

* Atrophic kidneys with maximum length<8cm on recent (<1 month) renal ultrasound, CT scan, or renal MRI
* High clinical suspicion of Complement-mediated aHUS (including familial history of aHUS)
* High clinical suspicion of typical HUS (including Shiga Toxin-producing E. Coli infection) or Thrombotic thrombocytopenic purpura
* High clinical suspicion of secondary HUS related to autoimmune disease (including lupus, scleroderma, antiphospholipid syndrome, ANCA vasculitis), or C3 glomerulopathy.
* High clinical suspicion of recent hemorrhagic or ischemic stroke.
* ADAMTS 13<10%, HIV or HCV infection, positivity of 2 markers among: anticardiolipin IgG/antiBeta2 GP1 IgG/lupus anticoagulant, positivity of ANCA (ELISA PR3 or MPO)
* Active infection
* Subjects with unresolved Neisseria meningitidis infection
* Subjects refusing Neisseria meningitidis vaccination or refusing antibioprophylaxis with oracillin (In case of penicillin allergy, antibioprophylaxis with macrolide couldbeproposed according to ANSM recommendations (azithromycin or roxithromycin)).
* Contra-indication to eculizumab or renin angiotensin system blockers
* Solid organ or haematopoietic transplant
* History (<1year) of active cancer or exposition to drugs associated with aHUS (< 3 months)
* Severe cognitive or psychiatric disorders, patients unable to give an informed consent.
* PCR SARS-CoV2 positive
* Pregnant or breastfeeding woman or ineffective contraception
* Persons deprived of their liberty by judicial or administrative decision,
* Persons under legal protection (guardianship, curatorship)
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2027-11-09 (Estimated)

PRIMARY OUTCOMES:
6-month response to therapy | 6 month
  6-month response to therapy, as defined by the absence of any of the following events: i) lack of renal efficacy at 6-month follow-up: persistent renal replacement therapy, eGFR <15ml/mn/1,73m2, or patient death; ii) lack of early hemolysis control with persistent hemolysis at W2 despite well conducted antihypertensive therapy. Any Eculizumab rescue in the control group will be considered as a failure.

SECONDARY OUTCOMES:
Frequency of Complement genetic rare variants | up to 12 months
Rate of renal replacement therapy | Week 13 and 12 months
  Evaluation of renal replacement therapy need at Week 13 and months 12
Frequency of severe infections | up to 12 months
  defined by the need for hospitalization
Time to resolution of hemolysis | up to 12 months
  Evaluation of hemolysis markers (anamia, thrombocytopenia, low hatoglobin, elevated lacticodehydrogenase, schistocytes)
Frequency of kidney lesions | up to 12 months
Costs relating to renal replacement therapy (or lack of) | up to 12 months
Costs relating to Eculizumab therapy | up to 12 months
Costs relating to other antihypertensive treatments | up to 12 months
Costs relating to hospitalizations | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tenon Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION